CLINICAL TRIAL: NCT04057248
Title: Digital Self-Management and Health Coaching for Type 2 Diabetes - Impact on Diabetes Clinical and Wellness Indicators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LabStyle Innovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CP-0010
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Results first posted 2021-03-30 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Digital platform and CDE coaching intervention for patients with type 2 Diabetes (Experimental): Patients provided with digital platform and connected devices. They undergo digital and human (CDE) intervention based on patient captured clinical data.
  Clinical parameters (HbA1C, weight, lipids profile, etc.) before and after intervention is assessed.
  Interventions: Device: Dario Blood Glucose Monitoring System; Behavioral: CDE

INTERVENTIONS:
Device: Dario Blood Glucose Monitoring System — Dario Blood Glucose Monitoring System (BGMS) with Dario App and Dario digital platform
Behavioral: CDE — Certified Diabetes Educator Sessions

SUMMARY:
Each subject enrolled in the study will be requested to complete an intake questionnaire including diabetes quality of life questions. The subject will use Dario Blood glucose monitoring system and will be contacted by a Certified Diabetes Educator (CDE) two to three times a month as well as have a direct communication using other communication channels such as mail, chat and text messaging (SMS) for lifestyle and diabetes management coaching for a total duration of three months. In the end of study, the subject will complete a diabetes quality of life questionnaire and have a blood test to evaluate its clinical parameters.

DETAILED DESCRIPTION:
This study is designed to assess the effect of digital self-monitoring platform used with the remote support of a Health coach on clinical outcomes and Diabetes quality of life.

Study design will be an open-label randomized trial of adults with Type 2. Patients are recruited through the Diabetes and Endocrinology Consultants center setting. Upon randomization to the intervention group, study participants will receive three months diabetes health coaching comprising of:

1. Two scheduled phone sessions with a Diabetes health coach a month;
2. Ongoing dual communication with the coach using digital communication channels such as chat, SMS and emails
3. Diabetes education, behavior modification, goal setting and reinforcement. The Dario App will record participant's glucose measurements and additional information captured by the patient such as medication intake, food and physical activity results.

The coach will get access to the patients' App captured information and will intervene ad necessary in the context of the clinical information.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, a subject must meet all the following criteria:

1. Adults 35 years of age or older
2. Diagnosed type 2 Diabetes
3. HbA1C test taken less than 2 months ago and is equal to or above 8.5%
4. Able to read, write and understand English
5. Have supported smartphone (see appendix C for the full smartphone list) with internet package for their service provider
6. The subject is able and agrees to sign the informed consent form

Exclusion Criteria:

1. Adults with impaired cognition
2. Cohabiting with a participant in the study
3. Have an underlying medical condition (such as kidney disease, hemoglobin variants, anemia) that may provide misleading A1C levels
4. Subject is critically ill
5. Subject has an impairment that prevents him/her from following the study procedures
6. Subject is not using medication that may interfere with the blood glucose measurement
7. HCT level which are outside Dario BGMS declared range (20%-60%)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Schorr, Dr., Principal Investigator — Diabetes and Endocrinology Consultants of Pennsylvania, LLC (Decpa LLC)
Locations (1):
- Diabetes and Endocrinology Consultants of Pennsylvania, LLC (Decpa LLC), Feasterville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant events occurred after study participant enrollment. 2 people were inactive.
Groups:
- Individual's Quality of Life and Clinical Parameters: Clinical parameters (HbA1C, weight, lipids profile, etc.)
  Dario Blood Glucose Monitoring System: Dario Blood Glucose Monitoring System (BGMS) with Dario App and Dario digital platform
  CDE: Certified Diabetes Educator Sessions
Period: Overall Study
Arm/Group | Individual's Quality of Life and Clinical Parameters
Started | 14
Completed | 12
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Individual's Quality of Life and Clinical Parameters
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
HBA1C>8.5 [Mean (Standard Deviation); unit: percentage of HBA1C in blood] — Population: 2 participants were inactive during the study
  percentage of HBA1C in blood
    number analyzed (Participants) | 12
    (all) | 10.2 (1.6)
Weight [Mean (Standard Deviation); unit: lbs] — Population: 2 participants were inactive during the study
  lbs
    number analyzed (Participants) | 12
    (all) | 233.9 (59.3)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Population: 2 participants were inactive during the study
  mg/dL
    number analyzed (Participants) | 12
    (all) | 180.3 (53.1)
Triglycerides value [Mean (Standard Deviation); unit: mg/dL] — Population: 2 participants were inactive during the study
  mg/dL
    number analyzed (Participants) | 12
    (all) | 192.5 (113.9)

OUTCOME MEASURES:

1. Primary Outcome: HbA1C Value at 3 Months From Subject Start of Study Compared to Baseline
Description: Change of HbA1C taken in blood test 3 month from the subject start of the study.
  Data was compared to baseline and reporting the HbA1C change from baseline measurement and 3 months after subject start of the clinical study.
  Measurement was conducted by Quest labs.
Time Frame: During 3 Months
Measure: Mean (Standard Deviation); unit: percentage of HBA1C in blood
Arm/Group | Individual's Quality of Life and Clinical Parameters
Number analyzed (Participants) | 12
percentage of HBA1C in blood | 8.2 (1.4)

2. Secondary Outcome: Cholesterol Value at 3 Months From Subject Start of Study
Description: Change of Cholesterol taken in blood test 3 month from the subject start of the study Data was compared to baseline and reporting the Cholesterol change from baseline measurement and 3 months after subject start of the clinical study.
  Measurement was conducted by Quest labs,
Time Frame: During 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Individual's Quality of Life and Clinical Parameters
Number analyzed (Participants) | 12
mg/dL | 179.0 (70.5)

3. Secondary Outcome: Weight Value at 3 Months From Subject Start of Study
Description: Change of Weight taken in the clinic at the beginning of the study and 3 month from the subject start of the study Data was compared to baseline and reporting the weight change from baseline measurement and 3 months after subject start of the clinical study.
Time Frame: During 3 months
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Individual's Quality of Life and Clinical Parameters
Number analyzed (Participants) | 12
lbs | 230.7 (58)

4. Secondary Outcome: Triglycerides Value at 3 Months From Subject Start of Study
Description: Change of Triglycerides taken in blood test 3 month from the subject start of the study Data was compared to baseline and reporting the Triglycerides change from baseline measurement and 3 months after subject start of the clinical study.
  Measurement was conducted by Quest labs,
Time Frame: During 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Individual's Quality of Life and Clinical Parameters
Number analyzed (Participants) | 12
mg/dL | 172.0 (121.5)

ADVERSE EVENTS:
Time Frame: 9 months
Description: Reporting requirements are provided in compliance with 21 CFR 812.150(b) (1).
  All-Cause Mortality: No mortalities were recorded during the study Serious Adverse Events: No serious adverse events were recorded during the study Other (Not Including Serious) Adverse Events: No other adverse events were recorded during the study
Arm/Group | Individual's Quality of Life and Clinical Parameters
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT04057248/Prot_SAP_000.pdf